CLINICAL TRIAL: NCT03661554
Title: BCMA Nano Antibody CAR-T Cells for the Treatment of Refractory Relapsed Multiple ,Single Center, Single Arm and Open Clinical Study of Myeloma
Brief Title: BCMA Nano Antibody CAR-T Cells for Patients With Refractory and Relapsed Multiple Myeloma
Acronym: BCMA CAR-T
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Pregene (ShenZhen) Biotechnology Company, Ltd. (Industry)
Collaborators: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG 1801
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: In this study, a 3 + 3 dose gradient climbing design was used. Three dosage groups, 5 x 106 / kg, 1 x 107 / kg and 1.5 x 107 / kg, were divided into three groups.
Masking Description: Clinical study of BCMA nano-antibody CAR-T cells in the treatment of refractory recurrent multiple myeloma (single center, single arm, open clinical study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): This clinical study, "BCMA nano-antibody CAR-T cells in the treatment of refractory recurrent multiple myeloma clinical research," is a single center, single arm, open design. The aim is to study the safety and efficacy of BCMA nano antibody CAR-T in the treatment of MM. In this study, a 3 + 3 dose gradient climbing design was used. Three dosage groups, 5x106 / kg, 1x107 / kg and 1.5x107 / kg, were divided into three groups.
  Interventions: Biological: BCMA CAR-T Cells

INTERVENTIONS:
Biological: BCMA CAR-T Cells — The Chinese name of CAR-T cells is chimeric antigen receptor T cells. It is through gene transfection technology, so that patients with T lymphocytes can carry B cell-specific antigens, so that T lymphocytes can selectively kill B lymphocyte-derived tumor cells.

SUMMARY:
This clinical study is an exploratory study, mainly to study the safety and efficacy of BCMA nano-antibody CAR-T in the treatment of MM. In this study, a 3 + 3 dose gradient climbing design was used. Three dosage groups, 5 x 106 / kg, 7.5 x 106 / kg and 1.5 x 107 / kg, were divided into three groups. Patients were enrolled in the sequence from low to high doses. When each dose group was completed, the next dose group could be enrolled if there was no more than 3-level toxicity or unpredictable severe toxicity. If the dose group had more than 3-level toxicity or unpredictable severe toxicity, two patients were enrolled to observe if there was any toxicity. Sexual occurrence, if two patients in each group developed grade 3 or more toxicity or unpredictable severe toxicity, the dose group was the dose-limiting group, and the dose group in front of the group was the maximum tolerated dose, at which the initial efficacy was observed. Nine patients were enrolled in the hill climbing test, and six patients were enrolled in the follow-up preliminary efficacy study, with an estimated 15 enrolled.

DETAILED DESCRIPTION:
The aim of this study is to study the safety and efficacy of BCMA nanoantibody CAR-T in the treatment of MM. BCMA CAR is composed of BCMA nano-antibody, CD8 strand region, transmembrane region and 4-1BB costimulatory domain, and CD3-_T cell activation domain. BCMA nano-antibody CAR-T cells were prepared by lentivirus infection of T cells. In this study, a 3 + 3 dose gradient climbing design was used. Three dosage groups, 5x106 / kg, 1x107 / kg and 1.5x107 / kg, were divided into three groups. Patients were enrolled in the sequence from low to high doses. When each dose group was completed, the next dose group could be enrolled if there was no more than 3-level toxicity or unpredictable severe toxicity. If the dose group had more than 3-level toxicity or unpredictable severe toxicity, two patients were enrolled to observe if there was any toxicity. Sexual occurrence, if two patients in each group developed grade 3 or more toxicity or unpredictable severe toxicity, the dose group was the dose-limiting group, and the dose group in front of the group was the maximum tolerated dose, at which the initial efficacy was observed. Nine patients were enrolled in the hill climbing test, and six patients were enrolled in the follow-up preliminary efficacy study, with an estimated 15 enrolled. After transfusion, adverse events were closely monitored and therapeutic effects were evaluated on the 28th day after transfusion. Follow-up was conducted every 6 weeks within 6 months and every 10 weeks after 6 months. To evaluate the safety and efficacy of BCMA nano antibody CAR-T in the treatment of refractory and relapsed MM.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, the expected survival time is greater than 3 months;
* Active MM was diagnosed, BCMA positive;
* At present, there is no effective treatment, such as chemotherapy or recurrence after hematopoietic stem cell transplantation, or patients voluntarily choose to infuse anti-BCMA nano-antibody CAR-T cells as the first treatment;
* ECOG : 0-2 points;
* Cardiac function: no heart disease or coronary heart disease, cardiac function 1-2;
* Liver function: TBIL < 3 ULN, AST < 2.5 ULN, ALT < 2.5 ULN;
* Renal function: Cr < 1.25 ULN;
* Patients with smooth peripheral venous access can meet the needs of intravenous drip;
* There are no other serious diseases (such as autoimmune diseases, immunodeficiency and organ transplantation) that are inconsistent with this protocol;
* There was no history of malignancy;
* Women of childbearing age must be tested for negative blood pregnancy tests within 7 days, and subjects of childbearing age must use appropriate contraceptive measures during the trial and within 3 months after the trial;
* Patients agreed to participate in the clinical study and signed the informed consent form.

Exclusion Criteria:

* Pregnant women or lactating women (women of childbearing age need to have a pregnancy check);
* Severe infectious diseases were found in the first 4 weeks of admission;
* Active hepatitis B or C viral hepatitis;
* HIV infected patients;
* Suffering from severe autoimmune or immunodeficiency diseases;
* Severe allergic constitution;
* Severe mental disorders;
* Systematic overuse of glucocorticoids within the first four weeks of admission (except for inhaled corticosteroids);
* Suffering from severe heart, liver, renal insufficiency, diabetes and other diseases;
* In the past 3 months, he participated in other clinical studies or previous treatment of other gene products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Any adverse events associated with BCMA nanoscale CAR-T cell therapy during the trial period

CONTACTS AND LOCATIONS:
Locations (1):
- Pregene Shenzhen Biotechnology Co., Ltd., Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided